CLINICAL TRIAL: NCT02181413
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind Study of Oral Ixazomib Citrate (MLN9708) Maintenance Therapy in Patients With Multiple Myeloma Following Autologous Stem Cell Transplant
Brief Title: A Study of Oral Ixazomib Citrate (MLN9708) Maintenance Therapy in Participants With Multiple Myeloma Following Autologous Stem Cell Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C16019; U1111-1155-8695 (Other: WHO); 2013-002076-41 (EudraCT Number); C16019CTIL (Registry Identifier: Israel MOH); NL.47795.029.14 (Registry Identifier: CCMO); 173116 (Registry Identifier: HC-CTD); 1036024001 (Registry Identifier: TCTIN); SNCTP000001745 (Registry Identifier: SNCTP)
Record Dates: First submitted 2014-06-27; First posted 2014-07-04 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma; Autologous Stem Cell Transplant
Keywords: Drug therapy; Ixazomib citrate
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Ixazomib citrate placebo-matching capsules, orally, once on Days 1, 8 and 15 in a 28-day cycle for Cycles 1 through 26 until PD, unacceptable toxicity, or discontinuation for alternate reasons.
  Interventions: Drug: Placebo
- Ixazomib Citrate (Experimental): Ixazomib citrate 3 mg, capsules, orally, once, on Days 1, 8 and 15 in a 28-day cycle for Cycles 1 through 4. Ixazomib citrate 4 mg, capsules, orally, once, on Days 1, 8 and 15 in a 28-day cycle for Cycles 5 through 26 until PD, unacceptable toxicity, or discontinuation for alternate reasons. Participants who have had any dose reductions due to adverse events (AEs) would not be dose escalated.
  Interventions: Drug: Ixazomib Citrate

INTERVENTIONS:
Drug: Ixazomib Citrate — Ixazomib citrate capsules
  Other Names: MLN9708
  Arms: Ixazomib Citrate
Drug: Placebo — Ixazomib citrate placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of ixazomib citrate maintenance therapy on progression-free survival (PFS), compared to placebo, in participants with newly diagnosed multiple myeloma (NDMM) who have had a response (complete response [CR], very good partial response [VGPR], or partial response [PR]) to induction therapy followed by high-dose therapy (HDT) and autologous stem cell transplant (ASCT).

DETAILED DESCRIPTION:
The investigational drug being tested in this study is called ixazomib citrate. Ixazomib citrate is being tested to slow disease progression and improve overall survival in people who have NDMM and who have had any type of positive response to induction therapy followed by HDT and ASCT. This study will look at the effect ixazomib citrate has on the length of time that participants are free of progressive disease (PD) and their overall survival (OS).

The study enrolled 656 participants. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need, or if the disease has progressed and the information is required for planning the next treatment):

* Ixazomib citrate 3 mg for the first 4 cycles, then 4 mg for the remaining 22 cycles
* Placebo (dummy inactive pill) - this is a capsule that looks like the study drug but has no active ingredient.

All participants will be asked to take one capsule on Days 1, 8 and 15 of each 28-day cycle, for up to 26 cycles (approximately 24 months).

This multi-center trial will be conducted globally. The overall time to participate in this study is up to 107 months. Participants will make 28 visits to the clinic during the treatment period and will continue to make visits after treatment has ended. During this initial follow up period, participants will be assessed for disease status with follow up every 12 weeks. After the next line of therapy begins, follow-up will occur every 12 weeks until death or termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female participants 18 years or older with a confirmed diagnosis of symptomatic multiple myeloma according to standard criteria.
2. Documented results of cytogenetics/ fluorescence in situ hybridization (FISH) obtained at any time before transplant, and International Staging System (ISS) staging at the time of diagnosis available.
3. Underwent standard of care (SOC) induction therapy (induction therapy must include proteasome inhibitor (PI) and/or immunomodulating drugs (IMiD)-based regimens as primary therapy for multiple myeloma), followed by a single autologous stem cell transplant (ASCT) with a high-dose melphalan (200 mg/m^2) conditioning regimen, within 12 months of diagnosis. Vincristine, Adriamycin [doxorubicin], and dexamethasone (VAD) is not an acceptable induction therapy for this trial.
4. Started screening no earlier than 75 days after transplant, completed screening within 15 days, and randomized no later than 115 days after transplant.
5. Must have not received post-ASCT consolidation therapy.
6. Documented response to ASCT (PR, VGPR, CR/stringent complete response [sCR]) according to IMWG criteria.
7. ECOG performance status of 0 to 2.
8. Female participants who:

   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 90 days after the last dose of study drug, AND
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.) Male participants, even if surgically sterilized (ie, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, AND
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
9. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
10. Suitable venous access for the study-required blood sampling.
11. Is willing and able to adhere to the study visit schedule and other protocol requirements.
12. Must meet the following clinical laboratory criteria at study entry:

    * Absolute neutrophil count (ANC) ≥ 1,000 per cubic milliliter (/mm^3) and platelet count ≥ 75,000/mm^3. Platelet transfusions to help participants meet eligibility criteria are not allowed within 3 days before randomization.
    * Total bilirubin ≤ 1.5 * the upper limit of the normal range (ULN).
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 * ULN.
    * Calculated creatinine clearance ≥ 30 milliliter per minute (mL/min).

Exclusion Criteria:

1. Multiple myeloma that has relapsed following primary therapy or is not responsive to primary therapy. For this study, stable disease following ASCT will be considered nonresponsive to primary therapy.
2. Double (tandem) ASCT.
3. Radiotherapy within 14 days before the first dose of study drug.
4. Diagnosed or treated for another malignancy within 5 years before randomization or previously diagnosed with another malignancy with evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
5. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period.
6. Major surgery within 14 days before randomization.
7. Central nervous system involvement.
8. Infection requiring intravenous (IV) antibiotic therapy or other serious infection within 14 days before randomization.
9. Diagnosis of Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
10. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
11. Systemic treatment with strong cytochrome P450 3A (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before randomization in the study.
12. Active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
13. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens (eg, peripheral neuropathy that is Grade 1 with pain or Grade 2 or higher of any cause).
14. Psychiatric illness/social situation that would limit compliance with study requirements.
15. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
16. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal (GI) procedure that could interfere with the oral absorption or tolerance of treatment.
17. Treatment with any investigational products within 60 days before the first dose of the study drug regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (227):
- United States (6):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - West Virginia University Hospital, Morgantown, West Virginia
- Argentina (6):
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Instituto de Hematologia Y Medicina Clinica Dr Ruben Davoli, Rosario, Santa Fe Province
  - Sanatorio Britanico de Rosario, Rosario, Santa Fe Province
  - Sanatorio Parque de Rosario, Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Iturraspe, Santa Fe
- Australia (9):
  - St George Hospital, Kogarah, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (4):
  - Elisabethinen Hospital Linz, Linz
  - Salzburger Landeskliniken, Salzburg
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Klinik Ottakring (fruher: Wilhelminenspital), Vienna
- Belgium (6):
  - Centre Hospitalier Jolimont-Lobbes, La Louvière, Hainaut
  - Centre Hospitalier Universitaire Ambroise Pare, Mons, Hainaut
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Sint-Jan AV, Bruges, West-Vlaanderen
  - ZNA Middelheim, Antwerp
  - ZNA Stuivenberg, Antwerp
- Brazil (15):
  - Hospital Das Clinicas Da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Instituto de Oncologia Do Parana, Curitiba, Paraná
  - Liga Paranaense de Combate Ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital de Clinicas de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Mae de Deus Center Hospital Giovanni Battista, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas, Florianópolis, Santa Catarina
  - Instituto Joinvilense de Hematologia E Oncologia, Joinville, Santa Catarina
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital de Base Da FAMERP, São José do Rio Preto, São Paulo
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Universidade Federal do Rio de Janeiro - UFRJ, Rio de Janeiro
  - Irmandade Da Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Canada (2):
  - University Health Network, Toronto, Ontario
  - MUHC-Glen Site, Montreal, Quebec
- Colombia (3):
  - Instituto Nacional de Cancerologia Colombia, Bogota, Cundinamarca
  - Fundacion Valle Del Lili, Cali, Valle del Cauca Department
  - Hospital Pablo Tobon Uribe, Medellín
- Czechia (6):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Kralovehradeck Kraj
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- Denmark (7):
  - Herlev Hospital, Herlev, Capital
  - Aalborg Universitetshospital, Aalborg, North Denmark
  - Aarhus Universitetshospital Arhus Sygehus, Aarhus N
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense
  - Sjallands Universitetshospital, Roskilde, Roskilde
  - Vejle Sygehus, Vejle
- France (5):
  - Hopital Antoine Beclere, Clamart, Hauts-de-Seine
  - Hotel Dieu - Nantes, Nantes, Loire-Atlantique
  - CHRU Lille, Lille, Nord
  - Hopital Universitaire Dupuytren, Limoges
  - Groupe Hospitalier Necker Enfants Malades, Paris
- Germany (23):
  - University Clinic Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum Mannheim Universitatsklinikum gGmbH, Mannheim, Baden-Wurttemberg
  - Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg
  - LMU Klinikum der Universitat Munchen, München, Bavaria
  - Universitatsklinikum Wurzburg, Würzburg, Bavaria
  - Klinikum Darmstadt GmbH, Darmstadt, Hesse
  - Klinikum Frankfurt Hochst GmbH, Frankfurt am Main, Hesse
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Universitatsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Uniklinik Koln, Cologne, North Rhine-Westphalia
  - Universitatsklinikum Essen, Essen, North Rhine-Westphalia
  - Evangelisches Krankenhaus Essen Werden gGmbH, Essen, North Rhine-Westphalia
  - Katholisches Krankenhaus Hagen gGmbH, Hagen, North Rhine-Westphalia
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz, Rhineland-Palatinate
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony
  - Helios Klinikum Berlin-Buch, Berlin
  - Charite - Universitatsmedizin Berlin, Berlin
  - Asklepios Klinik St. Georg, Hamburg
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - KRH Klinikum Siloah-Oststadt-Heidehaus, Hanover
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Universitatsklinikum Tubingen, Tübingen
- Greece (4):
  - Evangelismos General Hospital of Athens, Athens, Attica
  - Laiko General Hospital of Athens, Athens, Attica
  - Alexandra Hospital, Athens
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Del-pesti Centrumkorhaz- Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Israel (14):
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Centre, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center - PPDS, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center PPDS -, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center - PPDS, Petah Tikva
  - Sheba Medical Center - PPDS, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - ZIV Medical Center, Safed
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
  - Shamir Medical Center Assaf Harofeh, Tzrifin
- Italy (14):
  - Presidio Ospedaliero di Pescara, Pescara, Abruzzo
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Lombardy
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - IRCCS Centro Di Riferimento Oncologico Della Basilicata, Rionero in Vulture, Potenza
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Ancona, The Marches
  - Azienda Ospedaliera S Maria Di Terni, Terni, Umbria
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia - INCIPIT - PIN, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Az. Osp. Universitaria San Martino- IST, Genova
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l - PPDS, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda, Milan
  - Ospedale Infermi di Rimini, Rimini
- Japan (17):
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Saitama Medical Center, Kawagoe, Saitama
  - Juntendo University Hospital, Bunkyo, Tokyo
  - Chiba University Hospital, Chiba, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Nagoya City University Hospital, Nagoya
  - National Hospital Organaization Shibukawa Medical Center, Shibukawa
  - National Hospital Organization Disaster Medical Center, Tachikawa
  - Toyohashi Municipal Hospital, Toyohashi
- Mexico (2):
  - Centro de Investigacion Farmaceutica Especializada de Occidente, SC - PPDS, Guadalajara, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
- Netherlands (5):
  - VU Medisch Centrum, Amsterdam, North Holland
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Norway (4):
  - Vestre Viken HF Sykehuset Asker Og Barum, Gjelta, Oppland
  - St. Olav's University Hospital, Trondheim, Sor-Trondelag
  - Oslo Universitetssykehus HF, Ulleval, Oslo
  - Stavanger Universitetssykehus, Stavanger
- Poland (6):
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Wojskowy Instytut Medyczny, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów, Silesian Voivodeship
  - Szpital Specjalistyczny w Brzozowie, Brzozów
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
- Portugal (4):
  - Hospital de Braga, Braga
  - Centro Hospitalar E Universitario de Coimbra EPE, Coimbra
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto
  - Centro Hospitalar de Sao Joao, E.P.E., Porto
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital (SGH), Singapore
- South Africa (3):
  - Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Mary Potter Oncology Centre, Pretoria, Gauteng
  - Albert Alberts Stem Cell Transplant Centre, Pretoria, Gauteng
- South Korea (9):
  - National Cancer Center, Goyang, Gyeonggido
  - Chungnam National University Hospital, Daejeon
  - Gachon University Gil Medical Center Pharmacy, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (13):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid, Madrid, Communidad Delaware
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Clinic de Barcelona, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Institut Catala d'Oncologia Girona, Girona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario HM Sanchinarro CIOCC, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Asistencial Universitario de Salamanca H. Clinico, Salamanca
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- Sweden (5):
  - Helsingborg Lasarett, Helsingborg, Skåne County
  - Skanes Universitetssjukhus Lund, Lund, Skåne County
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Akademiska Sjukhuset I Uppsala, Uppsala
- Switzerland (2):
  - Universitatsspital Basel, Basel, Basel-Stadt (de)
  - Universitatsspital Zurich, Zurich, Zurich (de)
- Taiwan (5):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chang Gung Medical Foundation-Kaoshiung Branch, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation Chiayi Chang Gung Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Thailand (2):
  - Chulalongkorn University, Bangkok, Krung Thep Maha Nakhon-Bangkok
  - Phramongkutklao Hospital, Bangkok, Krung Thep Maha Nakhon-Bangkok
- Turkey (Türkiye) (7):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Ankara University Medical Faculty PPDS, Ankara
  - Pamukkale Universitesi Tip Fakultesi Hastanesi, Denizli
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
  - Karadeniz Technical University Faculty of Medicine, Trabzon
- MNPE Kyiv Center of Bone Marrow Transplantation of executive body of Kyiv council, Kyiv, Ukraine
- United Kingdom (11):
  - Southampton General Hospital, Southampton, Hampshire
  - Barts Health NHS Trust, Royal London Hospital, Ambrose King Centre, London, London, City of
  - Kings College Hospital, London, London, City of
  - Imperial College Healthcare NHS Trust, London, London, City of
  - Churchill Hospital, Oxford, Oxfordshire
  - Royal Marsden Hospital - Surrey, Sutton, Surrey
  - St James University Hospital, Leeds, Yorkshire
  - Royal Hallamshire Hospital, Sheffield, Yorkshire
  - University Hospitals Leicester, Leicester
  - University College London Hospitals (UCLH), London
  - Singleton Hospital - PPDS, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Paiva B, Manrique I, Dimopoulos MA, Gay F, Min CK, Zweegman S, Spicka I, Teipel R, Mateos MV, Giuliani N, Cavo M, Hopkins CR, Fu W, Suryanarayan K, Vorog A, Li C, Wang B, Estevam J, Labotka R, Dash AB. MRD dynamics during maintenance for improved prognostication of 1280 patients with myeloma in the TOURMALINE-MM3 and -MM4 trials. Blood. 2023 Feb 9;141(6):579-591. doi: 10.1182/blood.2022016782. PMID 36130300
- [Derived] Kaiser M, Beksac M, Gulbrandsen N, Schjesvold F, Hajek R, Moreau P, de Arriba de la Fuente F, Mateos MV, West S, Spencer A, Rajkumar SV, Suryanarayan K, Czorniak M, Li C, Teng Z, Labotka R, Dimopoulos MA. Adverse event management in the TOURMALINE-MM3 study of post-transplant ixazomib maintenance in multiple myeloma. Ann Hematol. 2020 Aug;99(8):1793-1804. doi: 10.1007/s00277-020-04149-5. Epub 2020 Jul 1. PMID 32613281
- [Derived] Schjesvold F, Goldschmidt H, Maisnar V, Spicka I, Abildgaard N, Rowlings P, Cain L, Romanus D, Suryanarayan K, Rajkumar V, Odom D, Gnanasakthy A, Dimopoulos M. Quality of life is maintained with ixazomib maintenance in post-transplant newly diagnosed multiple myeloma: The TOURMALINE-MM3 trial. Eur J Haematol. 2020 May;104(5):443-458. doi: 10.1111/ejh.13379. Epub 2020 Feb 22. PMID 31880006
- [Derived] Dimopoulos MA, Gay F, Schjesvold F, Beksac M, Hajek R, Weisel KC, Goldschmidt H, Maisnar V, Moreau P, Min CK, Pluta A, Chng WJ, Kaiser M, Zweegman S, Mateos MV, Spencer A, Iida S, Morgan G, Suryanarayan K, Teng Z, Skacel T, Palumbo A, Dash AB, Gupta N, Labotka R, Rajkumar SV; TOURMALINE-MM3 study group. Oral ixazomib maintenance following autologous stem cell transplantation (TOURMALINE-MM3): a double-blind, randomised, placebo-controlled phase 3 trial. Lancet. 2019 Jan 19;393(10168):253-264. doi: 10.1016/S0140-6736(18)33003-4. Epub 2018 Dec 10. PMID 30545780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 167 sites globally to take part in this study from 16 July 2014 to 8 September 2023.
Pre-assignment Details: Participants with newly diagnosed multiple myeloma (NDMM) who underwent induction therapy according to regional standard of care (SoC), followed by high-dose melphalan (200 milligrams per meter square [mg/m^2]) and Autologous Stem Cell Transplant (ASCT) were enrolled in a 3:2 ratio to receive ixazomib citrate or placebo.
Groups:
- Placebo: Ixazomib citrate placebo-matching capsules, orally, once on Days 1, 8 and 15 in a 28-day cycle for Cycles 1 through 26 until progressive disease (PD), unacceptable toxicity, or discontinuation for alternate reasons.
- Ixazomib Citrate: Ixazomib citrate 3 mg, capsules, orally, once, on Days 1, 8 and 15 in a 28-day cycle for Cycles 1 through 4. Ixazomib citrate 4 mg, capsules, orally, once, on Days 1, 8 and 15 in a 28-day cycle for Cycles 5 through 26 until PD, unacceptable toxicity, or discontinuation for alternate reasons. Participants who had any dose reductions due to adverse events (AEs) were not dose escalated.
Period: Overall Study
Arm/Group | Placebo | Ixazomib Citrate
Started | 261 | 395
Intent-to-Treat (ITT) Population | 261 | 395
Safety Population | 259 | 394
Per Protocol (PP) Population | 256 | 387
Completed | 206 | 322
Not Completed | 55 | 73
Not completed — Withdrawal by Subject | 45 | 61
Not completed — Reason Not Specified | 2 | 5
Not completed — Lost to Follow-up | 8 | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population was defined as all participants who were randomized and had post randomization data.
Groups:
- Ixazomib Citrate: Ixazomib citrate 3 mg, capsules, orally, once, on Days 1, 8 and 15 in a 28-day cycle for Cycles 1 through 4. Ixazomib citrate 4 mg, capsules, orally, once, on Days 1, 8 and 15 in a 28-day cycle for Cycles 5 through 26 until PD, unacceptable toxicity, or discontinuation for alternate reasons. Participants who had any dose reductions due to AEs were not dose escalated.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ixazomib Citrate | Total
Number analyzed (Participants) | 261 | 395 | 656
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (7.92) | 56.8 (8.17) | 57.4 (8.10)
Age, Customized [Count of Participants; unit: Participants]
  <60 years | 127 | 229 | 356
  ≥60 and <75 years | 134 | 166 | 300
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 143 | 242
  Male | 162 | 252 | 414
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 25
  Not Hispanic or Latino | 240 | 362 | 602
  Unknown or Not Reported | 10 | 19 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 213 | 315 | 528
  Black or African American | 3 | 7 | 10
  Asian | 36 | 59 | 95
  Other | 1 | 2 | 3
  Not Reported | 8 | 12 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 11 | 17 | 28
  Japan | 9 | 13 | 22
  Korea, Republic Of | 17 | 23 | 40
  Singapore | 4 | 8 | 12
  Taiwan, Province Of China | 3 | 10 | 13
  Thailand | 1 | 5 | 6
  Austria | 2 | 2 | 4
  Belgium | 5 | 5 | 10
  Czech Republic | 12 | 30 | 42
  Denmark | 11 | 20 | 31
  France | 7 | 11 | 18
  Germany | 26 | 50 | 76
  Greece | 22 | 38 | 60
  Hungary | 9 | 16 | 25
  Israel | 12 | 10 | 22
  Italy | 26 | 24 | 50
  Netherlands | 11 | 8 | 19
  Norway | 6 | 13 | 19
  Poland | 5 | 10 | 15
  Portugal | 2 | 8 | 10
  South Africa | 4 | 3 | 7
  Spain | 19 | 19 | 38
  Sweden | 4 | 7 | 11
  Switzerland | 3 | 0 | 3
  Turkey | 10 | 10 | 20
  Ukraine | 2 | 1 | 3
  United Kingdom | 14 | 21 | 35
  Argentina | 0 | 3 | 3
  Brazil | 3 | 5 | 8
  United States | 1 | 5 | 6
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with available height data.
  cm
    number analyzed (Participants) | 256 | 388 | 644
    (all) | 168.73 (10.347) | 169.71 (10.004) | 169.32 (10.145)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is the number of participants with available weight data.
  kg | 75.18 (14.648) | 75.93 (15.989) | 75.63 (15.463)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Population: Number analyzed is the number of participants with available BSA data.
  m^2
    number analyzed (Participants) | 256 | 388 | 644
    (all) | 1.87 (0.221) | 1.88 (0.235) | 1.88 (0.229)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of PD, as evaluated by an independent review committee (IRC) according to International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurred first. PD was defined as ≥25% increase from lowest value in: serum/urine M component; participants without measurable serum and urine M-protein levels, the difference between involved and uninvolved free light chain (FLC) levels must be >10 milligrams per deciliter (mg/dL); participants without measurable serum, urine M-protein levels and FLC levels, bone marrow plasma cell percent must have been ≥10%; new bone lesions/soft tissue plasmacytomas development/existing bone lesions/soft tissue plasmacytomas size increase; hypercalcemia development.
Time Frame: Randomization up to End of treatment (EOT) (24 months); thereafter followed up every 4 weeks (up to 45 months)
Population: Intent-to-Treat (ITT) population was defined as all participants who were randomized and had post randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 261 | 395
months | 21.3 [17.97 to 24.67] | 26.5 [23.69 to 33.81]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.002, Log Rank; P-value was based on log-rank test stratified by pre-induction regimen, International Staging System (ISS) stage and response after transplantation; Hazard Ratio (HR) = 0.720, 95% CI 2-sided [0.582 to 0.890] — HR was based on Cox's proportional hazard regression model stratified by pre-induction regimen, pre-induction ISS stage and response after transplantation. <1 HR indicates better prevention of progression in Ixazomib arm compared to Placebo

2. Secondary Outcome: Overall Survival (OS)
Description: OS was measured as the time from the date of randomization to the date of death.
Time Frame: Randomization up to end of follow up period (up to 107 months)
Population: ITT population was defined as all participants who were randomized and had post randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 261 | 395
months | NA [96.95 to NA] — Median and upper limit of 95% confidence interval (CI) were not estimable due to low number of participants with events. | NA [104.97 to NA] — Median and upper limit of 95% confidence interval (CI) were not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.850, Log Rank — P-value was based on log-rank test stratified by pre-induction regimen, ISS stage and response after transplantation; Hazard Ratio (HR) = 1.025, 95% CI 2-sided [0.789 to 1.332] — Hazard ratio is based on an unadjusted Cox's proportional hazard regression model stratified by induction regimen, pre-induction ISS, and response after transplantation, comparing the hazard rate of Ixazomib arm over the hazard rate of Placebo arm

3. Secondary Outcome: Percentage of Participants With Any Best Response Category Before PD or Subsequent Therapy
Description: Response was assessed according to IMWG criteria. Best response includes partial response (PR), very good partial response (VGPR) and complete response (CR). PR as per IMWG criteria is 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to less than (<)200 milligrams (mg) per 24 hours. VGPR is serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours. CR is negative immunofixation of serum and urine and disappearance of soft tissue plasmacytomas and <5% plasma cells in bone marrow. Stringent CR (sCR) is CR and normal FLC ratio and absence of clonal plasma cells (PCs) by immunohistochemistry or 2- to 4-color flow cytometry. The decimal values of percentages were subjected to rounding off.
Time Frame: Randomization up to EOT (up to 24 months) and thereafter every 4 weeks until initiation of the next line of therapy (up to 107 months)
Population: ITT population was defined as all participants who were randomized and had post randomization data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 261 | 395
percentage of participants
  PR | 10 | 12
  VGPR | 45 | 40
  CR | 42 | 44
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; CR; Test type: Superiority; p = 0.370, Cochran-Mantel-Haenszel — P-value is based on Cochran-Mantel-Haenszel (CMH) test stratified by pre-induction regimen, pre-induction international staging system (ISS), and response after transplantation at screening; Odds Ratio (OR) = 0.732, 95% CI 2-sided [0.365 to 1.466] — Odds ratio and CI are based on a logistic regression model with treatment group as a categorical predictor variable and pre-induction regimen, pre-induction ISS, and response after transplantation at screening as covariates

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the date of randomization to the date of first documentation of PD, using IMWG criteria. PD is defined as ≥25% increase from lowest value in: serum/urine M-component; participants without measurable serum and urine M-protein levels, the difference between involved and uninvolved FLC levels must be >10mg/dL; participants without measurable serum, urine M-protein levels and FLC levels, bone marrow plasma cell percent must be ≥10%;new bone lesions/soft tissue plasmacytomas development/existing bone lesions/soft tissue plasmacytomas size rise; hypercalcaemia development. Participants without documentation of PD at the time of analysis were censored at the date of last response assessment that is stable disease or better.
Time Frame: Randomization up to PD (up to 107 months)
Population: ITT Population was defined as all participants who were randomized and had post randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 261 | 395
months | 21.4 [18.10 to 24.67] | 26.6 [23.69 to 33.81]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.002, Log Rank — P-value was based on log-rank test stratified by pre-induction regimen, ISS stage and response after transplantation; Hazard Ratio (HR) = 0.716, 95% CI 2-sided [0.579 to 0.886] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Second Progression Free Survival (PFS2)
Description: PFS2 is defined as the time from the date of randomization to the date of objective disease progression on next line treatment or death from any cause (whichever occurs first). PD is defined as ≥25% increase from lowest value in: serum/urine M-component; participants without measurable serum and urine M-protein levels, the difference between involved and uninvolved FLC levels must be >10 mg/dL; participants without measurable serum, urine M-protein levels and FLC levels, bone marrow plasma cell percent must be ≥10%; new bone lesions/soft tissue plasmacytomas development/existing bone lesions/soft tissue plasmacytomas size rise; hypercalcaemia development.
Time Frame: Randomization up to EOT (24 months); thereafter followed up every 4 weeks until initiation of next-line therapy and then every 12 weeks until second progressive disease (PD2) or death (up to 107 months)
Population: ITT population was defined as all participants who were randomized and had post randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 261 | 395
months | 80.4 [68.7 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 84.0 [67.22 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.902, Log Rank — P-value was based on log-rank test stratified by pre-induction regimen, ISS stage and response after transplantation; Hazard Ratio (HR) = 1.015, 95% CI 2-sided [0.795 to 1.298] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Time to Start of the Next Line of Therapy
Description: Time to start of the next line of therapy was defined as the time from the date of randomization to the date of initiation dose of the next line of antineoplastic therapy following study treatment or death due to any cause, whichever occurred first. Participants who never took antineoplastic therapy were censored at the date of last contact or death.
Time Frame: Randomization up to 107 months
Population: ITT population was defined as all participants who were randomized and had post randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 261 | 395
months | 27.6 [24.48 to 31.61] | 33.1 [29.14 to 36.34]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.056, Log Rank; P-value was based on log-rank test stratified by pre-induction regimen, ISS stage and response after transplantation; Hazard Ratio (HR) = 0.833, 95% CI 2-sided [0.690 to 1.005] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Time to End of the Next Line of Therapy
Description: Time to end of the next line of therapy was defined as the time from the date of randomization to the date of last dose of the next line of antineoplastic therapy following study treatment or death due to any cause, whichever occurred first or date of last contact for participants who never took antineoplastic therapy.
Time Frame: Randomization up to 107 months
Population: ITT Population was defined as all participants who were randomized and had post randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 261 | 395
months | 50.4 [42.84 to 61.01] | 55.9 [49.61 to 61.86]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.431, Log Rank — P-value was based on log-rank test stratified by pre-induction regimen, ISS stage, and response after transplantation; Hazard Ratio (HR) = 0.922, 95% CI 2-sided [0.753 to 1.129] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Duration of the Next Line of Therapy
Description: Duration of the next line of therapy was defined as the time from the date of the first dose of the next line of therapy to the date of the last dose of the next antineoplastic therapy following study treatment or death due to any cause, whichever occurred first. Duration of the next line of therapy was analyzed on those participants who received the next line of therapy following the study treatment and duration was summarized using Kaplan-Meier method.
Time Frame: Up to 107 months
Population: ITT Population was defined as all participants who were randomized and had post randomization data. Overall number of participants analyzed indicates the number of participants who started next line of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 187 | 278
months | 12.3 [9.82 to 16.53] | 9.6 [7.49 to 12.06]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; Hazard Ratio (HR) = 1.179, 95% CI 2-sided [0.959 to 1.450] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Percentage of Participants Who Develop a New Primary Malignancy
Description: The decimal values of percentages were subjected to rounding off.
Time Frame: Up to 107 months
Population: Safety Population was defined as participants who received at least 1 dose of ixzaomib citrate or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 259 | 394
percentage of participants | 8 | 7

10. Secondary Outcome: Number of Participants With Conversion to Minimal Residual Disease (MRD) Negative
Description: MRD negativity (MRD-) is defined as absence of MRD and MRD positivity (MRD+) is defined as presence of MRD. The conversion rate from MRD positive to MRD negative was assessed and reported. Bone marrow aspirates and blood samples were sent to a central laboratory and were assessed for MRD using flow cytometry and a sequencing methodology.
Time Frame: Baseline up to EOT (up to 24 months)
Population: ITT population was defined as all participants who were randomized and had post randomization data. Overall number of participants analyzed indicates the number of participants with MRD+ at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 139 | 225
Participants | 27 | 39
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.814, Fisher Exact — P-value was based on Fisher's exact test comparing conversion to MRD- at any time post study entry between treatment groups

11. Secondary Outcome: Number of Participants With Maintenance of MRD Negativity
Description: MRD negativity is defined as absence of MRD and MRD positivity is defined as presence of MRD. The maintenance of MRD negativity up to the end of treatment was assessed and reported in participants converting from MRD+ at Baseline to MRD negative. Bone marrow aspirates and blood samples were sent to a central laboratory and were assessed for MRD using flow cytometry and a sequencing methodology.
Time Frame: Up to EOT (up to 24 months)
Population: ITT population was defined as all participants who were randomized and had post randomization data. Overall number analyzed is the number of participants who converted from MRD+ at Baseline to MRD negative.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 27 | 39
Participants | 25 | 37
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.805, Fisher Exact — [p-value comment as in outcome 10, analysis 1]

12. Secondary Outcome: Correlation Between MRD Status and Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the date of first documentation of PD as evaluated by an IRC according to IMWG criteria, or death due to any cause, whichever occurred first, assessed for up to 107 months in this outcome measure.
Time Frame: From randomization up to 107 months
Population: ITT population was defined as all participants who were randomized and had post randomization data. Overall number analyzed is the number of participants with data available for analyses. Number analyzed indicates the number of participants available for analysis in the specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 214 | 342
months
  MRD- at Study Entry: number analyzed (Participants) | 75 | 117
  MRD- at Study Entry | 32.5 [19.32 to NA] — Upper limit of 95% CI was not estimable due to censoring. | 38.6 [33.81 to NA] — Upper limit of 95% CI was not estimable due to censoring.
  MRD+ at Study Entry: number analyzed (Participants) | 139 | 225
  MRD+ at Study Entry | 18.5 [15.70 to 21.91] | 23.1 [20.24 to 25.69]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; MRD- at Study Entry; Test type: Superiority; p = 0.034, Log Rank — P-value was based on log-rank test stratified by pre-induction regimen, ISS stage and response after transplantation; Hazard Ratio (HR) = 0.612, 95% CI 2-sided [0.386 to 0.969] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixazomib Citrate; MRD+ at Study Entry; Test type: Superiority; p = 0.010, Log Rank — P-value was based on log-rank test stratified by pre-induction regimen, ISS stage and response after transplantation; Hazard Ratio (HR) = 0.704, 95% CI 2-sided [0.539 to 0.920] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Correlation Between MRD Status and Overall Survival (OS)
Description: OS was measured as the time from the date of randomization to the date of death, assessed for up to 107 months in this outcome measure.
Time Frame: From randomization up to 107 months
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 214 | 342
months
  MRD- at Study Entry: number analyzed (Participants) | 75 | 117
  MRD- at Study Entry | NA [84.90 to NA] — Median and upper limit of 95% CI were not estimable due to censoring. | NA [NA to NA] — Median, lower limit, and upper limit of 95% CI were not estimable due to censoring.
  MRD+ at Study Entry: number analyzed (Participants) | 139 | 225
  MRD+ at Study Entry | NA [90.74 to NA] — Median and upper limit of 95% CI were not estimable due to censoring. | 105.0 [91.47 to NA] — Upper limit of 95% CI was not estimable due to censoring.
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; MRD- at Study Entry; Test type: Superiority; p = 0.182, Log Rank — P-value was based on log-rank test stratified by pre-induction regimen, ISS stage and response after transplantation; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.414 to 1.184] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ixazomib Citrate; MRD+ at Study Entry; Test type: Superiority; p = 0.847, Log Rank — P-value was based on log-rank test stratified by pre-induction regimen, ISS stage and response after transplantation; Hazard Ratio (HR) = 0.966, 95% CI 2-sided [0.682 to 1.368] — [estimate comment as in outcome 2, analysis 1]

14. Secondary Outcome: OS Benefits in a High-Risk Population
Description: High-risk population included but was not limited to participants carrying deletion (del)17, t(4:14), t(14:16), amplification (ampl) 1q, del13, or del1p. OS was measured as the time from the date of randomization to the date of death.
Time Frame: Randomization up to 107 months
Population: ITT population was defined as all participants who were randomized and had post randomization data. Overall number analyzed is the number of participants present in the high-risk group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 54 | 61
months | 69.0 [33.25 to 92.98] | 64.2 [40.97 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.905, Log Rank — P-value was based on log-rank test stratified by pre-induction regimen, ISS stage and response after transplantation; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.583 to 1.613] — [estimate comment as in outcome 2, analysis 1]

15. Secondary Outcome: PFS Benefits in a High-Risk Population
Description: High-risk population included but not be limited to participants carrying deletion (del)17, t(4:14), t(14:16), amplification (ampl) 1q, del13, or del1p. PFS was defined as the time from the date of randomization to the date of first documentation of PD, as evaluated by an independent review committee according to IMWG criteria, or death due to any cause (whichever occurs first). PD is defined as ≥25% increase from lowest value in: serum/urine M-component; participants without measurable serum and urine M-protein levels, the difference between involved and uninvolved FLC levels must be >10mg/dL; participants without measurable serum, urine M-protein levels and FLC levels, bone marrow plasma cell percent must be ≥10%;new bone lesions/soft tissue plasmacytomas development/existing bone lesions/soft tissue plasmacytomas size rise; hypercalcaemia development.
Time Frame: Randomization up to 107 months
Population: ITT population was defined as all participants who were randomized and had post randomization data. Overall number of participants analyzed is the number of participants present in the high-risk group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 54 | 61
months | 16.8 [12.81 to 18.50] | 18.5 [12.06 to 31.15]

16. Secondary Outcome: Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status Score
Description: ECOG performance status assesses a participant's performance status on a 6-point scale ranging from 0=fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5=dead. Lower scores indicate improvement.
Time Frame: Baseline up to EOT (up to Month 24)
Population: Safety population was defined as participants who received at least 1 dose of ixazomib citrate or placebo. Overall number of participants analyzed indicates the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 252 | 371
score on a scale | 0.1 (0.63) | 0.0 (0.54)

17. Secondary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE) or Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation subject administered a drug. An AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. A TEAE was defined as an AE that started or worsened after first study drug administration and within 30 days of last dose of study drug. An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital abnormality or birth defect, an important medical event.
Time Frame: Up to 107 months
Population: Safety Population was defined as participants who received at least 1 dose of ixazomib citrate or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 259 | 394
Participants
  TEAEs | 241 | 382
  SAEs | 51 | 108

18. Secondary Outcome: Number of Participants With Markedly Abnormal Clinical Laboratory Values Reported as TEAEs
Description: Laboratory tests included chemistry, hematology and urinalysis. Abnormal laboratory value was assessed as an AE if the value led to discontinuation or delay in treatment, dose modification, therapeutic intervention, or was considered by the investigator to be a clinically significant change from baseline. A TEAE was defined as an AE that started or worsened after first study drug administration and within 30 days of last dose of study drug.
Time Frame: Up to 107 months
Population: Safety Population was defined as participants who received at least 1 dose of ixazomib citrate or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 259 | 394
Participants | 36 | 81

19. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Global Health Status/Quality of Life (GHS/QoL) Domain Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire used to assess the health-related quality of life of cancer patients. GHS/QoL domain is based on questions 29 ("How would you rate your overall health during the past week?") and 30 ("How would you rate your overall quality of life during the past week?") of the EORTC QLQ-C30 where the study participants' self-reported responses to the questions on a 7-point scale (1=very poor to 7=excellent). The raw GHS/QoL domain scores were linearly transformed to a scale ranging 0 (worse outcome) to 100 (best outcome), with higher scores indicating better quality of life. The change from baseline in EORTC QLQ-C30 GHS/QoL domain was evaluated by treatment group.
Time Frame: Baseline up to EOT (up to Month 24)
Population: ITT Population was defined as all participants who were randomized and had post randomization data. Overall number of participants analyzed indicates the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 237 | 349
score on a scale | -1.7 (1.57) | -4.1 (1.43)
Statistical Analysis 1: Comparison: Placebo vs Ixazomib Citrate; Test type: Superiority; p = 0.074, t-test, 2 sided; P-value was from the significance test for the coefficient of the interaction between treatment and visit; Least Squares (LS) Mean Difference = -2.3, 95% CI 2-sided [-4.9 to 0.2]

20. Secondary Outcome: Plasma Concentration of Ixazomib
Description: Plasma concentrations of the complete hydrolysis product of ixazomib citrate (ixazomib) were measured using a validated Liquid Chromatography-tandem Mass Spectrometry (LC/MS/MS) assay.
Time Frame: Day 1 of Cycle 1: 1 hour and 4 hours post-dose; Predose on Days 8 and 15 of Cycle 1, Days 1 and 8 of Cycle 2, Day 1 of Cycles 3 through 10 (each cycle length= 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as participants with at least one PK sample that was collected and analyzed. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Ixazomib Citrate
Number analyzed (Participants) | 393
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1: 1 Hour Post-dose: number analyzed (Participants) | 381
  Cycle 1 Day 1: 1 Hour Post-dose | 27.919 (24.7787)
  Cycle 1 Day 1: 4 Hours Post-dose: number analyzed (Participants) | 383
  Cycle 1 Day 1: 4 Hours Post-dose | 10.352 (9.8078)
  Cycle 1 Day 8: number analyzed (Participants) | 387
  Cycle 1 Day 8 | 1.584 (1.6707)
  Cycle 1 Day 15: number analyzed (Participants) | 382
  Cycle 1 Day 15 | 2.611 (1.4305)
  Cycle 2 Day 1: number analyzed (Participants) | 384
  Cycle 2 Day 1 | 1.946 (1.0984)
  Cycle 2 Day 8: number analyzed (Participants) | 374
  Cycle 2 Day 8 | 3.232 (2.0069)
  Cycle 3 Day 1: number analyzed (Participants) | 367
  Cycle 3 Day 1 | 2.258 (1.1508)
  Cycle 4 Day 1: number analyzed (Participants) | 367
  Cycle 4 Day 1 | 2.396 (1.7822)
  Cycle 5 Day 1: number analyzed (Participants) | 360
  Cycle 5 Day 1 | 2.400 (1.4921)
  Cycle 6 Day 1: number analyzed (Participants) | 350
  Cycle 6 Day 1 | 2.623 (1.6994)
  Cycle 7 Day 1: number analyzed (Participants) | 349
  Cycle 7 Day 1 | 2.691 (1.9842)
  Cycle 8 Day 1: number analyzed (Participants) | 338
  Cycle 8 Day 1 | 2.637 (1.7074)
  Cycle 9 Day 1: number analyzed (Participants) | 327
  Cycle 9 Day 1 | 2.610 (1.9380)
  Cycle 10 Day 1: number analyzed (Participants) | 321
  Cycle 10 Day 1 | 2.594 (1.9509)

21. Secondary Outcome: Time to Resolution of Peripheral Neuropathy (PN) Events
Description: Peripheral neuropathy is defined as the TEAE in the high-level term of peripheral neuropathies not elsewhere classified (NEC) according to Medical Dictionary for Regulatory Activities (MedDRA). A PN event is considered as improved if the event improves from the maximum grade. That is, all the grades recorded after the maximum grade is less than the maximum grade. Time to improvement is defined as the time from the initial onset date (inclusive) of the maximum grade to the first onset date that the toxicity grade is below the maximum grade with no higher grade thereafter, or the resolution date, whichever occurs first.
Time Frame: Up to 107 months
Population: Safety population was defined as participants who received at least 1 dose of ixazomib citrate or placebo. Overall number of participants analyzed indicates the number of participants with peripheral neuropathy events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 39 | 73
days | 159.0 [45.0 to 736.0] | 225.0 [117.0 to 421.0]

22. Secondary Outcome: Time to Improvement of PN Events
Description: PN is defined as the treatment-emergent adverse event in the high-level term of peripheral neuropathies not elsewhere classified (NEC) according to the Medical Dictionary for Regulatory Activities (MedDRA). A PN event is considered as resolved if its final outcome is resolved with no subsequent PN event of the same preferred term occurring on the resolution date or the day before and after. A PN event is considered as improved if the event improves from the maximum grade. That is, all the grades recorded after the maximum grade is less than the maximum grade. Time to improvement is defined as the time from the initial onset date (inclusive) of the maximum grade to the first onset date that the toxicity grade is below the maximum grade with no higher grade thereafter, or the resolution date, whichever occurs first.
Time Frame: Up to 107 months
Population: Safety population was defined as participants who received at least 1 dose of ixazomib citrate or placebo. Overall number of participants analyzed indicates number of participants with peripheral neuropathy events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Ixazomib Citrate
Number analyzed (Participants) | 39 | 73
days | 130.0 [36.0 to 520.0] | 134.0 [70.0 to 252.0]

ADVERSE EVENTS:
Time Frame: Randomization up to end of follow up period (107 months)
Description: All cause-mortality: ITT Population was defined as all participants who were randomized and had post randomization data. Serious and Other Adverse Events: Safety Population was defined as participants who received at least 1 dose of ixazomib citrate or placebo.
Arm/Group | Placebo | Ixazomib Citrate
All-Cause Mortality (participants affected / at risk) | 93/261 | 144/395
Serious Adverse Events (participants affected / at risk) | 51/259 | 108/394
Other Adverse Events (participants affected / at risk) | 229/259 | 371/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | Ixazomib Citrate (N=394)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atypical pneumonia (Infections and infestations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bacterial infection (Infections and infestations) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 3
C-reactive protein increased (Investigations) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Diplopia (Eye disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 4
Herpes zoster disseminated (Infections and infestations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Influenza (Infections and infestations) | 1 | 4
Influenza B virus test positive (Investigations) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Light chain analysis increased (Investigations) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 3
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2
Metapneumovirus infection (Infections and infestations) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 3
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pain (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 4
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Picornavirus infection (Infections and infestations) | 0 | 1
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 10 | 25
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 5
Radicular pain (Nervous system disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Varicella (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | Ixazomib Citrate (N=394)
Anaemia (Blood and lymphatic system disorders) | 8 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 | 105
Asthenia (General disorders) | 17 | 30
Back pain (Musculoskeletal and connective tissue disorders) | 47 | 77
Bone pain (Musculoskeletal and connective tissue disorders) | 19 | 37
Bronchitis (Infections and infestations) | 19 | 40
Conjunctivitis (Infections and infestations) | 10 | 28
Constipation (Gastrointestinal disorders) | 21 | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 87
Decreased appetite (Metabolism and nutrition disorders) | 17 | 21
Diarrhoea (Gastrointestinal disorders) | 61 | 135
Dizziness (Nervous system disorders) | 18 | 33
Dyspepsia (Gastrointestinal disorders) | 15 | 13
Fatigue (General disorders) | 43 | 79
Headache (Nervous system disorders) | 23 | 43
Herpes zoster (Infections and infestations) | 14 | 37
Hypertension (Vascular disorders) | 19 | 21
Influenza (Infections and infestations) | 29 | 38
Influenza like illness (General disorders) | 18 | 37
Insomnia (Psychiatric disorders) | 12 | 31
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 35
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 15 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 22
Nasopharyngitis (Infections and infestations) | 69 | 91
Nausea (Gastrointestinal disorders) | 40 | 154
Neuropathy peripheral (Nervous system disorders) | 19 | 40
Neutropenia (Blood and lymphatic system disorders) | 15 | 24
Oedema peripheral (General disorders) | 11 | 34
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 29
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 32
Paraesthesia (Nervous system disorders) | 8 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 23 | 41
Pharyngitis (Infections and infestations) | 9 | 20
Pneumonia (Infections and infestations) | 15 | 24
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 35
Pyrexia (General disorders) | 37 | 78
Rash macular (Skin and subcutaneous tissue disorders) | 8 | 24
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 24
Sinusitis (Infections and infestations) | 6 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 40
Upper respiratory tract infection (Infections and infestations) | 54 | 100
Vomiting (Gastrointestinal disorders) | 28 | 105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT02181413/Prot_002.pdf
  • Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT02181413/SAP_000.pdf